CLINICAL TRIAL: NCT01350674
Title: Role of EBUS-TBNA (Endobronchial Ultrasound Transbronchial Needle Aspiration- in Diagnosing Tuberculosis in Mediastinal and/or Hilar Lymph Nodes
Brief Title: Role of EBUS-TBNA in Diagnosing TB in Mediastinal/Hilar Lymph Nodes
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B07620109427; AK/10-10-3949/67 (Other: ethical committee UMC St Pieter Brussel Belgium)
Record Dates: First submitted 2011-04-28; First posted 2011-05-10 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2017-10

CONDITIONS: Tuberculosis
Keywords: mediastinal tuberculosis; endoscopy; EBUS; tuberculous lymphadenopathy; endobronchial ultrasound
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Lymph Node

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EBUS (Experimental): patients undergoing EBUS
  Interventions: Procedure: EBUS-TBNA

INTERVENTIONS:
Procedure: EBUS-TBNA — endobronchial ultrasound transbronchial needle aspiration

SUMMARY:
This is an observational prospective study. Role of EBUS-TBNA (endobronchial ultrasound transbronchial needle aspiration) is evaluated to diagnose tuberculosis in mediastinal and/or hilar lymph nodes.

The investigators analyse the specificity and sensibility of this technique to diagnose tuberculosis in mediastinal and/or hilar lymph nodes.

Patients with mediastinal and/or hilar lymph nodes on X-ray or CT thorax where a tuberculosis is the most probable cause and who have no parenchymal lesions suspected for tuberculosis and without other lymph nodes that are more easily accessible or palpable will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* patients with enlarged mediastinal and/or hilar lymph nodes on chest CT highly suspicious of tuberculosis (suggestive clinical history, suggestive echographic findings ...) without pulmonary lesions suspicious for tuberculosis or in whom the first evaluation with sputum examination, classical bronchoscopy, induced sputum didn't result in any diagnosis.
* patients aged 18 years or older
* patients need to sign the consent form after reading the information form

Exclusion Criteria:

* synchronic pulmonary lesions suspicious for tuberculosis or already proven tuberculosis by microscopic exam, PCR-technique and/or culture
* other affected ganglionary sites more easily accessible (cervical, supraclavicular, axillary ... region)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-12; Primary Completion 2017-12 (Actual); Study Completion 2018-03

PRIMARY OUTCOMES:
The ratio of tuberculosis in mediastinal lymph nodes | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Inge M Muylle, MD, Principal Investigator — CHU St. Pierre Brussels
Locations (1):
- CHU St. Pierre; pulmonology department, Brussels, Belgium